CLINICAL TRIAL: NCT05109520
Title: Evaluation of Glycemic Control and Quality of Life in Adults With Type 1 Diabetes During Continuous Glucose Monitoring When Switching to Insulin Glargine 300 U/mL: A FUTURE Substudy
Brief Title: Evaluation of Glycemic Control and Quality of Life in Adults With Type 1 Diabetes During Continuous Glucose Monitoring When Switching to Insulin Glargine 300 U/mL
Acronym: FUTURE-GLARE
Status: Completed | Type: Observational
Sponsor: prof dr Pieter Gillard (Other)
Collaborators: University Hospital, Antwerp (Other); Onze Lieve Vrouw Hospital (Other)
Responsible Party: Sponsor-Investigator, prof dr Pieter Gillard, Principal Investigators, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Other Study IDs: S65399
Record Dates: First submitted 2021-10-14; First posted 2021-11-05 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Glargine 300 U/mL; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- investigational group: Participants of the FUTURE study who switched during the study to Gla-300
  Interventions: Drug: Insulin Glargine 300 UNT/ML [Toujeo]
- control group: Participants of the FUTURE study who did not switch to Insulin Gla-300

INTERVENTIONS:
Drug: Insulin Glargine 300 UNT/ML [Toujeo] — Switch during standard routine care to Gla-300.
  Groups: investigational group

SUMMARY:
Retrospective multicenter study analyzing data gathered during the FUTURE study (S59342) to assess the effect of using Insulin Glargine 300 U/mL (Gla-300) on measures of diabetes control and quality of life.

Of the FUTURE participants, data about the type of insulin the participants used will be gathered. On the basis of these data participants will be divided in two groups (control or investigational).

Change in glycemic control and quality of life from before to after the switch to Gla-300 (investigational group) will be compared to the change of glycemic control and quality of life of the FUTURE participants who did not switch to Gla-300 (control group).

The FUTURE study was a 24-month during multicenter observational cohort study analyzing data on the use of the Abbott Freestyle Libre in people with diabetes. Data were gathered during standard clinical follow-up, and from questionnaires that were presented to the participants at defined time points.

ELIGIBILITY:
1. Investigational group

   Inclusion Criteria:
   * participant in the FUTURE study
   * diagnosed with type 1 diabetes ≥3 months before start of the FUTURE study
   * use of insulin pens for the entirety of the FUTURE study
   * used Insulin Detemir (Levemir®), Insulin Glargine 100 U/mL (Lantus®) or an equivalent as basal insulin before switch to Gla-300 (Toujeo®)
   * switched to Gla-300 (Toujeo®) during the FUTURE study for a sufficient amount of time (at least two consecutive diabetes consultations = 8 months)

   Exclusion Criteria:
   * use of Fast-acting insulin aspart (Fiasp®) before or after switch to Gla-300
   * not using bolus insulin (only basal insulin)
   * for women: pregnant or planning pregnancy during the FUTURE study
2. Control group

Inclusion Criteria:

* participant in the FUTURE study for at least 18 months
* diagnosed with type 1 diabetes ≥3 months before start of the FUTURE study
* use of insulin pens for the entirety of the FUTURE study
* use Insulin Detemir (Levemir®), Insulin Glargine 100 U/mL (Lantus®) or an equivalent as basal insulin during the entirety of the FUTURE study

Exclusion Criteria:

* use of Fast-acting insulin aspart (Fiasp®)
* not using bolus insulin (only basal insulin)
* for women: pregnant or planning pregnancy during the FUTURE study
* switch to Gla-300 (Toujeo®) or Insulin Degludec (Tresiba®) before 18 months in FUTURE study (if switched after 18 months, only data up to switch to Gla-300 [Toujeo®] or Insulin Degludec [Tresiba®] will be used for this control participant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with type 1 diabetes who participated in the FUTURE study.
Sampling Method: Non-Probability Sample
Enrollment: 867 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Time in range (TIR, 70-180 mg/dL) | maximum 24 months
  The difference in evolution of TIR (70-180 mg/dL, averaged per month) over 24 hours since switch to Gla-300

SECONDARY OUTCOMES:
HbA1c | maximum 24 months
  difference in HbA1c
Time in range (TIR, 70-180 mg/dL) | maximum 24 months
  difference in TIR (70-180 mg/dL, averaged per month) from 6 am to 10 pm, and from 10 pm to 6 am
Hypoglycemia | maximum 24 months
  difference in time in hypoglycemia (<54 mg/dL, <70 mg/dL, ≥54-<70 mg/dL; averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am
Hyperglycemia | maximum 24 months
  difference in time in hyperglycemia (>180 mg/dL, >250 mg/dL, >180-≤250 mg/dL; averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am
Mean glycemia | maximum 24 months
  difference in mean glucose (averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am
Glycemic variability | maximum 24 months
  difference in glycemic variability (standard deviation, coefficient of variation; averaged per month) over 24 hours, from 6 am to 10 pm, and from 10 pm to 6 am
Quality of life measured by the Short Form Health Survey 36-item (SF-36) version 2 questionnaire | maximum 24 months
  Quality of life measured by the Short Form Health Survey 36-item (SF-36) version 2 questionnaire (scale: 0 (low quality of life) - 100 (high quality of life))
Fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, worry | maximum 24 months
  Fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, worry (scale: 0 (not worried) - 72 (very worried))
Distress due to diabetes measured by the Problem Areas In Diabetes survey, short form (PAID-SF) questionnaire | maximum 24 months
  Distress due to diabetes measured by the Problem Areas In Diabetes survey, short form (PAID-SF) questionnaire (scale: 0 (no distress) - 20 (very distressed))
Treatment satisfaction measured by the Diabetes Treatment Satisfaction Questionnaire, status (DTSQs) | maximum 24 months
  Treatment satisfaction measured by the Diabetes Treatment Satisfaction Questionnaire, status (DTSQs) (scale: 0 (low satisfaction) - 36 (high satisfaction))

OTHER OUTCOMES:
Insulin dose | maximum 24 months
  difference in insulin dose (basal, bolus and total)
Body mass index | maximum 24 months
  difference in body mass index (BMI)
Severe hypoglycemia rate | maximum 24 months
  difference in self-reported severe hypoglycemic events
Hypoglycemic coma rate | maximum 24 months
  difference in self-reported hypoglycemic comas
Hospitalization | maximum 24 months
  difference in hospitalizations due to hypoglycemia or ketoacidosis

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Gillard, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (3):
- Belgium (3):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitaire Ziekenhuizen Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be shared upon a genuine request.

REFERENCES:
- [Derived] Charleer S, Fieuws S, De Block C, Bolsens N, Nobels F, Mikkelsen K, Mathieu C, Gillard P. Evaluation of Glucose Metrics in Adults with Type 1 Diabetes Switching to Insulin Glargine 300 U/mL: A Retrospective, Propensity-Score Matched Study. Diabetes Technol Ther. 2024 Jul;26(7):488-493. doi: 10.1089/dia.2023.0371. Epub 2024 Mar 6. PMID 38386438